CLINICAL TRIAL: NCT01787266
Title: Symptoms and Function During and After Pregnancy
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Britt Stuge, PT, PhD, Oslo University Hospital
Other Study IDs: PGQ2013; 129/12-303.0 (Other Grant/Funding Number: The Norwegian FONDET)
Record Dates: First submitted 2013-01-31; First posted 2013-02-08 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Pelvic Girdle Pain
MeSH Terms: conditions — Pelvic Girdle Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: pregnant women

SUMMARY:
The purpose of this study is to:

1. describe degree of symptoms and disability during and after pregnancy
2. to examine if women with pelvic girdle pain are able to correctly mark their pain location on a pain drawing
3. to examine the responsiveness of The Pelvic Girdle Questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy week 32-36
* Understand and read/write a questionnaire in Norwegian or English

Exclusion Criteria:

* Not able to understand and fill in a questionnaire

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant women in week 32 - 36
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
the pelvic girdle questionnaire | 10 weeks postpartum

SECONDARY OUTCOMES:
Pain intensity, Numeric rating scale | 10 weeks postpartum

OTHER OUTCOMES:
Short Form -8 (SF-8) | 10 weeks postpartum

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway